CLINICAL TRIAL: NCT05178030
Title: Validation of Mutation Analysis in Circulating Tumor DNA With a ddPCR Assay as Diagnostic and Follow-up Tool for Patients With a KIT Exon 11 Mutated GIST: GALLOP-11
Brief Title: The GALLOP-11 Study
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: 201900781
Record Dates: First submitted 2021-05-04; First posted 2022-01-05 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Gastro-intestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample and/or biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GALLOP-11: Patients with a proven KIT exon 11 mutated GIST covered by our in-house designed ddPCR assay.
  Interventions: Other: vena punction

INTERVENTIONS:
Other: vena punction — Regular 3-12 monthly follow-up by CT-scan will be compared to results of ctDNA analysis. Blood for analysis of mutation in ctDNA will be collected at the same moment a CT-scan is performed

SUMMARY:
An observational, multicenter study will be performed. Regular 3-12 monthly follow-up by CT-scan will be compared to results of ctDNA analysis. Blood for analysis of mutation in ctDNA will be collected at the same moment a CT-scan is performed. All samples will be analyzed at the reference Pathology laboratory at the UMCG. A part of the samples will also be analyzed in other institutions to implement the ddPCR. Primary endpoint is concordance between CT-scan and ctDNA analysis results, from which the negative predictive value (NPV) of our ddPCR assay will be calculated.

DETAILED DESCRIPTION:
This is an observational, non-interventional, multicenter study. The study will be performed within the Dutch GIST consortium (NKI-AvL, Erasmus MC, Radboud UMC, LUMC and UMCG). Patients diagnosed with GIST with a KIT exon 11 mutations that can be detected by our ddPCR assay are eligible. In this way we will study a homogenous patient population with GIST that (usually) responds very well to initial TKI treatment. Therefore, the KIT mutation status must be known. Patients can enter the study at any time point of their disease trajectory. Patients included in GALLOP-11 will have follow-up as described in the European Society of Medical Oncology and Dutch guidelines but with blood draws for ctDNA assessment at similar time points.

The primary objective is the negative predictive value (NPV) of the ddPCR assay result in relation to the results of the CT-scan and/or MRI scan (according to RECIST 1.1) at the same time point. Concordance of these results will be determined, from which the negative predictive value (NPV) of our ddPCR assay will be calculated. This is considered the most important value, as the most harmful scenario would be to miss progressive disease because not seen on ctDNA while it could have been seen on CT (and/or MRI). That would mean that ctDNA analysis is not reliable enough to replace CT-scan (and/or MRI) follow-up in the future.

To determine the negative predictive value, at least 250 patients need to have an evaluable follow-up strategy. To pursue a solid follow-up period within an achievable timeline, patients with at least four ctDNA measurements, accompanied by a CT-scan (and/or MRI scan), will be considered evaluable for the NPV analysis. Patients who have progression within four scans are always evaluable, since a positive outcome outweighs negative outcomes because it is known that ctDNA should have had measured change once it is seen on CT-scans (and/or MRI scans).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with GIST with a biopsy confirmed primary KIT exon 11 mutation covered by our KIT exon 11 ddPCR assay (mutation/deletion within target sequence of c.1665_1736);
2. Patients with an indication for at least 4 CT-scans concomitant with regular laboratory examination in a neoadjuvant, adjuvant and/or palliative care trajectory within the time frame of the study;
3. Age ≥18 years;
4. Written informed consent provided.

Exclusion Criteria:

1. Patients who are unable to comply with study procedures and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in a group of KIT exon 11 detectable (by our ddPCR assay) mutated GIST patients treated according to national guidelines. Newly diagnosed patients will be asked to participate as well as patients that are already on treatment. Furthermore, all GALLOP study patients that have a KIT exon 11 mutation that can be detected by our assay can participate.
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The negative predictive value of the ddPCR assay with regard to KIT exon 11 circulating tumour mutation | 3 years
  The negative predictive value of the ddPCR assay with regard to KIT exon 11 circulating tumour mutation digital droplet PCR (ddPCR) assay in relation to CT-scans.

SECONDARY OUTCOMES:
The sensitivity and specificity of the designed KIT exon 11 mutation | 3 years
  To establish the sensitivity and specificity of the designed KIT exon 11 mutation ddPCR assay
Technical validity of the ddPCR assay | 3 years
  The detection of ctDNA expressed in copies/mL and fractional abundance, assessed by the designed KIT exon 11 circulating tumour mutation digital droplet PCR (ddPCR) assay, in different laboratories, and by Agena Bioscience, will be assessed.
Clinical validity of the ddPCR assay | 3 years
  The first detection of increase in the level of the primary KIT exon 11 mutation in ctDNA determined in time to progression seen on standard radiological evaluation by CT-scan based on RECIST 1.1
Development of new assays to detect secondary mutations | 3 years
  Based on mutation analysis of tumor biopsies of patients with progressive disease, ctDNA assays will be designed and tested
Determination of time between first detection of secondary mutations and progression | 3 years
  Based on progression of disease on CT, we will analyze ctDNA of patients to determine wether secondary mutations could be found before radiologic progression

CONTACTS AND LOCATIONS:
Overall Officials: An KL Reyners, MD, PhD, Principal Investigator — Principal Investigator
Locations (5):
- Netherlands (5):
  - Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen
  - LUMC, Leiden
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam